CLINICAL TRIAL: NCT00312533
Title: Outcome Following Hylan F- 20 (Synvisc) + Corticosteroid Injections for the Treatment of Osteoarthritis of the Knee
Status: Completed | Type: Observational
Sponsor: Steadman Hawkins Research Foundation (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Other Study IDs: SHRF2006-01
Record Dates: First submitted 2006-04-06; First posted 2006-04-10 (Estimated); Last update posted 2008-08-25 (Estimated); Status verified 2008-08

CONDITIONS: Osteoarthritis, Knee
Keywords: knee; injection; function; osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Drug: Hylan F- 20

SUMMARY:
The goal of viscosupplementation is to replenish synovial fluid, which will improve patient symptoms and mobility. Viscosupplementation of the knee with hyaluronic acid injections has been shown to improve symptoms in patients with osteoarthritis. Recent studies have shown that this improvement may be highly variable based on the time from treatment, especially in the first 12 weeks following treatment. The purpose of this study is to document the outcomes following a treatment protocol in which corticosteroid is used in addition to the initial Synvisc injection in the series of three injections.

DETAILED DESCRIPTION:
Upon initial visit, all study patients will complete an informed consent. After consent, patients will complete the baseline questionnaire packet, which includes a questionnaire with several validated scoring systems. Following injection, patients will receive a diary to document any adverse events between the first and second injection. In one week, patients will return for a second visit to receive the second injection. Again they will be asked to maintain their diary of adverse events following the second injection. The patient will then receive the final injection at week 3 and will again complete a diary of events for one week. At 1 week, 3 weeks, 6 weeks, 12 weeks, and 26 weeks following the completed series of injections, the patients will complete a form that will include the pain, stiffness, and physical function subscales of the WOMAC score and a 10 point patient satisfaction question.

At 6 months, the patients will receive by mail the same questionnaire packet they received at baseline, with the addition of patient satisfaction and subsequent injury/treatment questions.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 to 80 years
* with a diagnosis of osteoarthritis of the knee. Diagnosis will be based on radiographic examination (Kellgren-Lawrence 2 or 3) or by previous arthroscopic diagnosis.

Surgical treatment for osteoarthritis will be limited to arthroscopic surgeries that include removal of loose bodies, resection of unstable meniscus tears and loose or unstable chondral flaps, removal of osteophytes if they limit extension, and lysis of adhesions. These types of treatments may provide symptomatic relief by increasing joint volume in knees with osteoarthritis and relieving joint contact pressures.

Exclusion Criteria:

* Patients with grade 4 Kellgren-Lawrence on radiographic examination will be excluded.
* Patients with a prior synovectomy on knee to be injected will be excluded.
* Patients will be excluded if they have rheumatoid disease or any other serious systemic disease, acute synovitis or excessive effusion, allergy to avian products/hyaluronan-based injection components/corticosteroid injection, pregnant, previous arthroscopic surgery within the last 6 months or had a joint infection within the previous 3 months.
* Patients who have undergone a prior synovectomy will not be included.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-04; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John R Steadman, MD, Principal Investigator — Steadman Hawkins Research Foundation
Locations (1):
- Steadman Hawkins Clinic, Vail, Colorado, United States